CLINICAL TRIAL: NCT02437591
Title: Open Label Study to Evaluate the Pharmacokinetics of Fidaxomicin in Inflammatory Bowel Disease (IBD) Subjects With Clostridium Difficile Infection (CDI)
Brief Title: Study to Evaluate the Pharmacokinetics of Fidaxomicin in Inflammatory Bowel Disease (IBD) Subjects With Clostridium Difficile Infection (CDI)
Acronym: PROFILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2819-MA-1003; 2014-003002-32 (EudraCT Number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Disease (IBD); Clostridium Difficile Infection (CDI)
Keywords: ASP2819; PAR-101; OPT-80; Inflammatory Bowel Disease (IBD); Clostridium difficile Infection (CDI); fidaxomicin; Dificlir
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections | interventions — Fidaxomicin; OPT 80

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fidaxomicin (Experimental): tablet twice daily
  Interventions: Drug: fidaxomicin

INTERVENTIONS:
Drug: fidaxomicin — oral
  Other Names: PAR-101; OPT-80; Dificlir; ASP2819

SUMMARY:
The purpose of this study is to investigate the plasma pharmacokinetics (PK) of fidaxomicin (FDX) and primary metabolite OP-1118 in Subjects with Inflammatory Bowel Disease (IBD) and C. difficile Infection (CDI).

This study will also compare CDI clinical response to the microbiological response in terms of magnitude of reduction of C. difficile total viable count and spore count during treatment with FDX and if achieved; the time to microbial eradication; determine time to negative CDI toxin assay in stool specimens during treatment with FDX; assess the stool concentrations of FDX and metabolite OP-1118 throughout therapy; assess the length of hospital stay, readmissions and resource utilization for IBD patients receiving FDX; record the incidence and severity of Adverse Events (AEs) and document the impact of treatment on Quality of Life as measured by the changes in Short Inflammatory Bowel Disease Questionnaire (IBDQ) score.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis or history of IBD for at least 3 months
* Subject has have active IBD defined by :

  * partial MAYO score (ulcerative colitis subjects) of 2 or more, where at least 1 point has to originate from blood in stool
  * Harvey-Bradshaw Index (HBI) (Crohn's disease subjects) of 5 or more, excluding points for complications
* CDI confirmed positive according to local standard testing for the presence of C. difficile within 48 hr prior to enrollment
* Female subject is not breastfeeding at Screening or while participating in this study
* Subject agrees to practice effective birth control from Screening and while participating in this study
* Subject agrees not to participate in another interventional study while participating in this study
* Male partner agrees not to donate sperm starting at screening and throughout the investigational period.

Exclusion Criteria:

* Subject has received more than one day of dosing of any CDI therapy within the 48 hrs prior to enrollment
* Subject is unable to swallow oral study medication
* Presence of an ostomy or short bowel syndrome
* Subject has a current diagnosis of toxic megacolon
* Subject is not willing to adhere to the provisions of treatment and observation specified in the protocol
* Subject has been enrolled into this study previously, has taken any investigational drug within 28 days or 5 half-lives, whichever is longer, prior to enrollment, or is currently participating in another clinical study which may influence the assessment of efficacy and/or safety endpoints of this study, in the opinion of the Sponsor
* Subject has previously participated in a CDI vaccine study
* Subject has hypersensitivity to FDX or any of its components
* Subject has a condition which, in the Investigator's opinion, makes the Subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of fidaxomicin: Maximum plasma concentration (Cmax) | Day 1, Day 5 and Day 10
Pharmacokinetic parameter of OP-1118: Maximum plasma concentration (Cmax) | Day 1, Day 5 and Day 10
Pharmacokinetic parameter of fidaxomicin: Area under the curve from 0 to 12 hrs (AUC12) | Day 1
Pharmacokinetic parameter of OP-1118: Area under the curve from 0 to 12 hrs (AUC12) | Day 1
Pharmacokinetic parameter of fidaxomicin and OP-1118: Metabolite to Parent Ratio (MPR) | Day 1
Pharmacokinetic parameter of fidaxomicin: Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau) | Day 5 and Day 10
Pharmacokinetic parameter of OP-1118: Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau) | Day 5 and Day 10
Pharmacokinetic parameter of fidaxomicin: The time after dosing when Cmax occurs (tmax) | Day 1, Day 5 and Day 10
Pharmacokinetic parameter of OP-1118: The time after dosing when Cmax occurs (tmax) | Day 1, Day 5 and Day 10
Pharmacokinetic parameter of fidaxomicin: Apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F) | Day 5 and Day 10
Pharmacokinetic parameter of OP-1118: Apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F) | Day 5 and Day 10
Pharmacokinetic parameter of fidaxomicin: Concentration immediately prior to dosing at multiple dosing (Ctrough) | Day 5 and Day 10
Pharmacokinetic parameter of OP-1118: Concentration immediately prior to dosing at multiple dosing (Ctrough) | Day 5 and Day 10

SECONDARY OUTCOMES:
CDI clinical response | Day 12
Microbiological response of C. difficile total viable count, spore count, microbiological eradication and negative CDI toxin assay | Day 5 and Day 10
Stool concentrations of fidaxomicin and its metabolite OP-1118 | Day 1, Day 5 and Day 10
Length of hospital stay, readmissions and resource utilization | up to Day 180
Safety as assessed by incidence and severity of adverse events | up to Day 180
Health related quality of life as assessed by short IBDQ score | Day 10, Day 26, Day 40, Day 90 and Day 180
  Inflammatory Bowel Disease Questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe Ltd.
Locations (12):
- Site AT43001, Graz, Austria
- France (2):
  - Site FR33002, Clichy
  - Site FR33001, Paris
- Site GR30004, Athens, Greece
- Italy (2):
  - Site IT39003, Padua
  - Site IT39001, Roma
- Poland (2):
  - Site PL48002, Warsaw
  - Site PL48003, Warsaw
- Russia (3):
  - Site RU70003, Moscow
  - Site RU70002, Moscow
  - Site RU70001, Saint Petersburg
- Site GB44002, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Hogenauer C, Mahida Y, Stallmach A, Marteau P, Rydzewska G, Ivashkin V, Gargalianos-Kakolyris P, Michon I, Adomakoh N, Georgopali A, Tretter R, Karas A, Reinisch W. Pharmacokinetics and safety of fidaxomicin in patients with inflammatory bowel disease and Clostridium difficile infection: an open-label Phase IIIb/IV study (PROFILE). J Antimicrob Chemother. 2018 Dec 1;73(12):3430-3441. doi: 10.1093/jac/dky368. PMID 30260412
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=227